CLINICAL TRIAL: NCT07187440
Title: A Prospective, Multi-center, Observational Study to Evaluate the Clinical Outcomes of Agalsidase Alfa Enzyme Replacement Therapy Among Chinese Patients With Fabry Disease in Real-world Clinical Practice
Brief Title: A Study of Agalsidase Alfa Enyzme Replacement Therapy in Chinese Children and Adults With Fabry Disease
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-675-4013
Record Dates: First submitted 2025-09-18; First posted 2025-09-23 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Fabry Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants with Fabry disease will receive enzyme replacement therapy (ERT) with agalsidase alfa under routine clinical practice settings.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is a non-interventional study

SUMMARY:
Fabry Disease is a rare blood disorder that some people are born with. People with Fabry disease have low levels of an enzyme called alpha-galactosidase A. This enzyme helps to cut down fat-like substances. Without alpha-galactosidase A, large forms of these substances build up and clot in blood vessels. Over time, this can affect vital organs (especially the heart, kidneys, and brain) causing serious health problems with advancing age. Agalsidase alfa (Replagal®) is a human enzyme made in the laboratory and may provide higher levels of alpha-galactosidase A. Replagal® works the same way as natural alpha-galactosidase A does.

The main aim of this study is to learn more about the treatment with Replagal® in Chinese children and adults with Fabry disease. The study aims to assess the heart and kidney function in people with Fabry disease who are routinely treated with Replagal®. Other aims are to learn about the change in heart and kidney function, impact on quality of life, how the treatment with Replagal® works for people with Fabry Disease, and how safe the treatment with Replagal® is in routine real-world settings.

Participants will receive with Replagal® per the routine treatment settings in China. No study-specific visits to the clinical are scheduled.

ELIGIBILITY:
Inclusion Criteria

Participants who meet all of the following criteria are eligible for this study:

* Participant is greater than or equal to (>= 7) years old.
* Participant with confirmed diagnosis of Fabry disease (by investigator).
* Participant never received or has received ERT (agalsidase alfa or agalsidase beta) within 12 weeks at most prior to enrolment.
* Participant who will receive ERT with agalsidase alfa in routine clinical practice settings.
* For >= 18 years old, participant should sign the informed consent form (ICF); for 8-17 years old, participant and his (her) parents/ legally authorized representative (LAR) should both sign the ICF; for < 8 years old, participant will give assent and his (her) parents/legally authorized representative should sign the ICF accordingly.

Exclusion Criteria

* Participant will be excluded if they have documented New York Heart Association (NYHA) functional Class IV heart failure symptoms (Implantable cardioverter-defibrillator [ICD] implanted excluded), third-degree atrioventricular block (ICD implanted excluded), acute myocardial infarction within the last 3 months and severe stroke (NIH Stroke Scale [NIHSS] >= to 21).
* Participant has enrolled in Fabry disease interventional clinical trial currently.
* Other situations that the investigator considers not suitable for participation in this study.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with Fabry disease who receive ERT with agalsidase alfa in routine clinical practice settings in China.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Annualized Rate of Change in Left Ventricular Mass Index (LVMI) | Up to 18 months
  The annualized rate of change in LVMI will be estimated using linear mixed effects model.
Annualized Rate of Change in Estimated Glomerular Filtration Rate (eGFR) | Up to 18 months

SECONDARY OUTCOMES:
Annualized Rate of Change in Left Ventricular Posterior Wall Dimensions (LVPWD) | Up to 18 months
Annualized Rate of Change in Ejection Fraction (EF) | Up to 18 months
Change From Baseline Over Time in LVMI | Baseline, up to 18 months
Change From Baseline Over Time in LVPWD | Baseline, up to 18 months
Change From Baseline Over Time in EF | Baseline, up to 18 months
Annualized Rate of Change in Urinary Albumin to Creatinine Ratio (UACR) | Up to 18 months
Annualized Rate of Change in Urine Protein Creatine Ratio (UPCR) | Up to 18 months
Change From Baseline Over Time in eGFR | Baseline, up to 18 months
Change From Baseline Over Time in UACR | Baseline, up to 18 months
Change From Baseline Over Time in UPCR | Baseline, up to 18 months
Change From Baseline Over Time in 24-hour (h) Urine Protein | Baseline, up to 18 months
Change From Baseline Over Time in 36-Item Short Form Health Survey (SF-36) | Baseline, up to 18 months
  SF-36 is a questionnaire that evaluates a person's HRQOL. SF-36 includes 36 questions related to 8 health dimensions: physical functioning, role-physical (role limitations due to physical health problems), bodily pain, general health, vitality (energy/fatigue), social functioning, role-emotional (role limitations due to emotional problems), and mental health. Based on these 4 scales (physical functioning, role-physical, bodily pain, general health), the physical component summary (PCS) score is generated which ranges between 0 and 100, with higher scores indicating a better quality of life. A positive change from Baseline indicates improvement.
Change From Baseline Over Time in Mainz Severity Score Index (MSSI) | Baseline, up to 18 months
  MSSI is an instrument for quantifying the overall severity of the signs and symptoms of Fabry disease. The MSSI assigns scores based on the presence and severity of signs and symptoms in four areas: general, neurologic, cardiovascular, and renal. Each of the signs and symptoms is weighted in accordance with its relationship to morbidity.
  MSSI scoring ranges from 0 (healthy) to 76 (maximum severity), and it is divided into severity bands of mild (<20), moderate (20-40), and severe (>40) affliction. Higher score indicates more severity.
Number of Participants With Clinically Significant Adverse Events (AEs) With Agalsidase Alfa Treatment | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (18):
- China (18):
  - The First Affiliated Hospital Of USTC (AnHui Provincial Hospital), Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Fuzhou University Provincial Affiliated Hospital, Fuzhou, Fujian
  - The Second Affiliated Hospital ZheJiang University School Of Medicine, Hangzhou, Guangdong
  - ShanTou Central Hospital, Shantou, Guangdong
  - The University Of Hong Kong-ShenZhen Hospital, Shenzhen, Guangdong
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - The First Affiliated Hospital With NanJing Medical University(JiangSu Province Hospital), Nanjing, Jiangsu
  - The First Affiliated Hospital Of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi 'an Jiaotong University, Xi'an, Shaanxi
  - Second Hospital Of ShanXi Medical University, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - TianJin Chest Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/